CLINICAL TRIAL: NCT02062268
Title: Study of KAP and Influential Factors on Drink Driving in Public in Jiangsu Province in China
Brief Title: The Study of KAP on Drink Driving in Jiangsu Province in China
Acronym: KAP
Status: Completed | Type: Observational
Sponsor: Jiangsu Province Centers for Disease Control and Prevention (Network)
Responsible Party: Sponsor
Other Study IDs: jsdd1301
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2016-09-01 (Estimated); Status verified 2014-02

CONDITIONS: Drink Driving
Keywords: KAP; drink driving; public; Jiangsu province; China
MeSH Terms: conditions — Driving Under the Influence

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Urban area in South Jiangsu Province: health education & law enforcement
  Interventions: Behavioral: health education & law enforcement
- urban area in Middle Jiangsu Province: health education & law enforcement
  Interventions: Behavioral: health education & law enforcement
- urban area in North Jiangsu Province: health education & law enforcement
  Interventions: Behavioral: health education & law enforcement
- rural area in South Jiangsu Province: health education & law enforcement
  Interventions: Behavioral: health education & law enforcement
- rural area in North Jiangsu Province: health education & law enforcement
  Interventions: Behavioral: health education & law enforcement

INTERVENTIONS:
Behavioral: health education & law enforcement

SUMMARY:
Conduct a KAP survey before and after intervention and describe the current knowledge, attitudes and behaviors on drink driving in public and analyse the influential factors to provide rational strategies to enhance the awareness on drink driving in public.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-70, resident for more than 6 months.

Exclusion Criteria:

* less than 18 or older than 70, or provisional resident.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: urban and rural residents in Jiangsu province aged 18-70.
Sampling Method: Probability Sample
Enrollment: 3565 (Actual)
Dates: Start 2014-03; Primary Completion 2015-01 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
self-report drink driving rate in public decreases by 2.5% | one and a half year

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoning LI, MD, Study Director — Jiangsu CDPC
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China